CLINICAL TRIAL: NCT00767117
Title: A Phase I, Open-label, Randomized Cross-over, 2-period, 2-way Interaction Trial to Investigate the Pharmacokinetic Interaction Between Lopinavir/Ritonavir and TMC125 Both at Steady-state in Healthy Subjects.
Brief Title: TMC125-TiDP2-C197: A Phase I Trial to Investigate the Pharmacokinetic Interaction Between Lopinavir/Ritonavir and TMC125 Both at Steady-state in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015526
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-05

CONDITIONS: HIV
Keywords: TMC125-C197; TMC125-TiDP2-C197; HIV; DDI; Lopinavir; Intelence; Kaletra; Ritonavir; Etravirine; Interaction; Pharmacokinetics; Steady-state
MeSH Terms: interventions — etravirine; Lopinavir; Ritonavir

INTERVENTIONS:
Drug: Etravirine; Lopinavir; Ritonavir

SUMMARY:
The purpose of the study is to determine the effect of steady-state concentrations of LPV, co-administered with a low dose of ritonavir, on the steady-state pharmacokinetics of TMC125 and to determine the effect of steady-state concentrations of TMC125 on the steady-state pharmacokinetics of LPV, co-administered with a low dose of ritonavir.

DETAILED DESCRIPTION:
This is a Phase I, open-label, randomized (patients are assigned different treatments based on chance), 2-period, 2-way cross-over interaction trial to investigate the pharmacokinetic interaction (study of the bodily absorption, distribution, metabolism, and excretion of drugs) between lopinavir/ritonavir (LPV/rtv) and TMC125, both at steady-state.The trial population will consist of 16 healthy volunteers. In 2 consecutive sessions, healthy volunteers will receive Treatment A and Treatment B, in a randomized sequence. In Treatment A, 200 mg TMC125 b.i.d.will be administered for 7 days (from Day 1 to Day 7) with an additional morning dose on Day 8. In Treatment B, 400/100 mgLPV/rtv twice a day will be administered for 15 days (from Day 1 to Day15) with an additional morning dose on Day 16, while 200 mgTMC125 b.i.d. will be co-administered from Day 9 to Day 15 with an additional morning dose on Day 16. Subsequent sessions will be separated by a washout period of at least 2 weeks. Full pharmacokinetic profiles of TMC125 will be determined over the 12-hour dosing interval after the morning intake on Day 8 of Treatment A and on Day 16 of Treatment B. Full pharmacokinetic profiles of LPV and ritonavir will be determined over the 12-hour dosing interval after the morning intake on Days 8 and 16 of Treatment B. All treatments will be administered under fed conditions and will be taken within 10 minutes after a meal. Safety and tolerability evaluations will be recorded continuously. Treatment A = 200 mg TMC125 b.i.d. will be administered for 7 days (from Day 1 to Day 7) with an additional morning dose on Day 8. Treatment B = 400/100 mg LPV/rtv b.i.d. will be administered for 15 days (from Day 1 to Day 15) with an additional morning dose on Day 16, while 200 mg TMC125 b.i.d. will be co-administered from Day 9 to Day 15 with an additional morning dose on Day 16.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* Normal weight as defined by a Quetelet Index (Body Mass Index [BMI], weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form (ICF) signed voluntarily before the first trial-related activity
* Able to comply with protocol requirements
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram (ECG), vital signs, and the results of blood biochemistry, hematology and a urinalysis carried out at screening.

Exclusion Criteria:

* No positive HIV-1 or HIV-2 test at Screening
* No hepatitis A infection (confirmed by hepatitis A antibody IgM), or hepatitis B infection (confirmed by hepatitis B surface antigen), or hepatitis C infection (confirmed by hepatitis C virus antibody) at study screening
* No currently active or underlying gastro-intestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease
* No currently significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability
* No history of significant skin disease such as, but not limited to, rash or eruptions, drug allergies, food allergies, dermatitis, eczema, psoriasis, or urticaria
* No previously demonstrated clinically significant allergy or hypersensitivity to any of the excipients of the investigational medication administered in this trial
* No use of concomitant medication, including over-the-counter products and dietary supplements. Over-the-counter systemic medication must have been discontinued at least 7 days prior to the first dose of study medication
* prescribed medication and all products containing Hypericum perforatum must have been discontinued at least 14 days before the first dose of study medication, except for paracetamol/acetaminophen and ibuprofen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determine the effect of steady-state concentrations of LPV/low dose ritonavir, on the steady-state pharmacokinetics of TMC125 and vice versa.

SECONDARY OUTCOMES:
Evaluate the short-term safety and tolerability of the concomitant use of TMC125 and LPV, co-administered with low-dose ritonavir in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- See also: A Phase I, open label, randomized, cross-over, 2-period, 2-way interaction trial to investigate the pharmacokinetic interaction between lopinavir/ritonavir and TMC125 both at steady-state in healthy subjects. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1016&filename=CR015526_CSR.pdf